CLINICAL TRIAL: NCT01525706
Title: EUS Guided Ethanol With Paclitaxel Ablation for Pancreatic Mucinous Cystic Neoplasm
Brief Title: Endoscopic Ultrasound (EUS) Guided Ethanol With Paclitaxel Ablation for Pancreatic Mucinous Cystic Neoplasm
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: University of Western Ontario, Canada (Other)
Responsible Party: Principal Investigator, Brian Yan, Assistant Professor of Medicine, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UWO18494
Record Dates: First submitted 2012-02-01; First posted 2012-02-03 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Mucinous Cystic Tumor With Moderate Dysplasia; Mucinous Cystadenoma of Pancreas; Mucinous Cystadenocarcinoma of Pancreas; Benign Neoplasm of Pancreas
Keywords: Endoscopic Ultrasound; Pancreatic Mucinous Cystic Neoplasm; Fine Needle Injection; Ethanol Ablation; Paclitaxel Ablation
MeSH Terms: interventions — Ethanol; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ethanol and Paclitaxel Injection (Experimental): All patients will receive at least one treatment with alcohol and paclitaxel.
  Interventions: Drug: Ethanol and Paclitaxel Injection

INTERVENTIONS:
Drug: Ethanol and Paclitaxel Injection — Endoscopic ultrasound will be used to locate and assess the pancreatic cyst. The fluid contents will be aspirated using a fine needle and sent for tumor marker analysis and cytology. With the needle maintained in the same position, 99% ethanol will be injected into the cyst. After 3-5 minutes of lavage, the entire volume of fluid will be removed from the cyst. The same volume of paclitaxel minus 1 mL [3mg/ml diluted in normal saline from original concentration of 6mg/mL] will be injected and left in the cyst. The needle is then retracted and the procedure completed. Patients will receive oral prophylactic antibiotics for 5 days after the procedure. Clinical follow up with MRI imaging with be done at 6, 12, 18, and 24 months. For those with a persistent cyst at 12 months, a repeat EUS FNI procedure will be done.
  Other Names: Ethanol; Paclitaxel

SUMMARY:
Pancreatic cysts are becoming diagnosed more frequently due to the increased use and sensitivity of imaging. A subset of these cysts are pre-cancerous, therefore suggested treatment is surgery for removal. However, surgery involves significant risks and emerging opinion suggests that not all cysts need to be surgically removed. An alternative therapy would be ideal, in particular for those where surgical risk outweighs the benefits of resection. Ethanol and paclitaxel ablation of pancreatic cysts may be a viable alternative to surgical resection.

Our hypothesis is that ethanol with paclitaxel ablation is a safe and effective method for treatment in those with per-cancerous, mucinous pancreatic cysts.

ELIGIBILITY:
Inclusion Criteria:

1. Mucinous cystic neoplasm defined by cyst fluid analysis [23, 28]:

   * CEA > 192ng/mL
   * Amylase < 800 IU/L
   * Cytology negative for malignant cells
   * No communication of cyst with pancreatic duct on 2 imaging studies (EUS, CT, MRCP, or ERCP)
2. Cyst size > 15mm but <50mm
3. 3 or fewer cyst compartments
4. Age ≥18 and ≤ 85

Exclusion Criteria:

1. Inability to safely undergo EUS examination with standard conscious sedation
2. Inability for safe FNA needle insertion into the cyst (eg: intervening vessel)
3. Inability to undergo MRI (metal implants/cardiac pacemaker/defibrillator, claustrophobia)
4. Coagulopathy (INR>1.5 or platelets<50)
5. Active pancreatitis or pancreatic infection
6. Active sepsis/bacteremia
7. Inability to provide informed consent
8. Pregnancy
9. Breastfeeding women

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-09; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Efficacy: Cyst Resolution | 6 months
  Proportion of patients without cysts at 6 months
Efficacy: Degree of Ablation | 6 months
  Degree of cyst epithelial ablation in those undergoing resection

SECONDARY OUTCOMES:
Safety | 30 day
  Safety of ethanol/paclitaxel ablation
Efficacy: Change of tumor markers | 12 month
  Change of CEA level in those with persistent/recurrent cyst
Efficacy: Cyst Resolution | 12 month
  Proportion of patients without cysts at 12 months
Efficacy: Cyst Resolution | 18 months
  Proportion of patients without cysts at 18 months
Efficacy: Cyst Resolution | 24 months
  Proportion of patients with no cysts at 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Yan, MD, FRCPC, Principal Investigator — Western University, Canada
Locations (1):
- St. Joseph's Health Care, London, Ontario, Canada

REFERENCES:
- [Result] Oh HC, Seo DW, Song TJ, Moon SH, Park DH, Soo Lee S, Lee SK, Kim MH, Kim J. Endoscopic ultrasonography-guided ethanol lavage with paclitaxel injection treats patients with pancreatic cysts. Gastroenterology. 2011 Jan;140(1):172-9. doi: 10.1053/j.gastro.2010.10.001. Epub 2010 Oct 13. PMID 20950614
- [Result] Oh HC, Seo DW, Lee TY, Kim JY, Lee SS, Lee SK, Kim MH. New treatment for cystic tumors of the pancreas: EUS-guided ethanol lavage with paclitaxel injection. Gastrointest Endosc. 2008 Apr;67(4):636-42. doi: 10.1016/j.gie.2007.09.038. Epub 2008 Feb 11. PMID 18262182
- [Result] DeWitt J, DiMaio CJ, Brugge WR. Long-term follow-up of pancreatic cysts that resolve radiologically after EUS-guided ethanol ablation. Gastrointest Endosc. 2010 Oct;72(4):862-6. doi: 10.1016/j.gie.2010.02.039. PMID 20883866
- [Result] DeWitt J, McGreevy K, Schmidt CM, Brugge WR. EUS-guided ethanol versus saline solution lavage for pancreatic cysts: a randomized, double-blind study. Gastrointest Endosc. 2009 Oct;70(4):710-23. doi: 10.1016/j.gie.2009.03.1173. Epub 2009 Jul 4. PMID 19577745